CLINICAL TRIAL: NCT03100851
Title: Effect of Fermented Milk Containing Lactobacillus Casei Strain Shirota on Chinese People With Constipation
Brief Title: Effect of Probiotic on Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Agricultural University (Other)
Responsible Party: Principal Investigator, Fazheng Ren, Professor, China Agricultural University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUConstipation-01
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

ARMS (1):
- LcS intervention (Experimental): Patients with constipation received dietary supplement with Lactobacaiilus casei strain Shirota.
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei strain Shirota — a bottle of 100 mililiter probiotic dairy beverage containing 10^8 CFU Lactobacillus casei strain Shirota every day after lunch.

SUMMARY:
Constipation is a prevalent intestinal disorder. Lactobacillus casei strain Shirota (LcS) shows potential effect on alleviating constipation. This study evaluated the impact of fermented milk containing LcS on stool consistency and frequency. The stool short chain fatty acid and gut microbiota were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* meet ROME Ⅲ criteria for functional constipation
* normal body mass index between 18.5 and 29.9

Exclusion Criteria:

* had a serious disease;
* used systemic antibiotics or antimycotics medication and antidiarrheal or laxative medication in the 30 days prior to the study;
* allergic to milk protein;
* constipated because of organic or neurological lesions;
* participated in any other studies within 2 months prior to this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-08-02 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
change of stool consistency | change from baseline stool consistency at four-week intervention
change of defecation frequency | change from baseline defecation frequency at four-week intervention
change of constipation-related symptom scores | change from baseline constipation-related symptom scores at four-week intervention

SECONDARY OUTCOMES:
Changes in stool short chain fatty acid content | change from baseline stool short chain fatty acid content at four-week intervention
Changes in gut microbiota | change from baseline gut microbiota at four-week intervention

REFERENCES:
- [Background] Chu H, Zhong L, Li H, Zhang X, Zhang J, Hou X. Epidemiology characteristics of constipation for general population, pediatric population, and elderly population in china. Gastroenterol Res Pract. 2014;2014:532734. doi: 10.1155/2014/532734. Epub 2014 Oct 16. PMID 25386187
- [Background] Sandler RS, Drossman DA. Bowel habits in young adults not seeking health care. Dig Dis Sci. 1987 Aug;32(8):841-5. doi: 10.1007/BF01296706. PMID 3608732
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Tigchelaar EF, Bonder MJ, Jankipersadsing SA, Fu J, Wijmenga C, Zhernakova A. Gut microbiota composition associated with stool consistency. Gut. 2016 Mar;65(3):540-2. doi: 10.1136/gutjnl-2015-310328. Epub 2015 Aug 14. No abstract available. PMID 26276682
- [Background] Khalif IL, Quigley EM, Konovitch EA, Maximova ID. Alterations in the colonic flora and intestinal permeability and evidence of immune activation in chronic constipation. Dig Liver Dis. 2005 Nov;37(11):838-49. doi: 10.1016/j.dld.2005.06.008. Epub 2005 Oct 5. PMID 16169298
- [Background] Husebye E, Hellstrom PM, Sundler F, Chen J, Midtvedt T. Influence of microbial species on small intestinal myoelectric activity and transit in germ-free rats. Am J Physiol Gastrointest Liver Physiol. 2001 Mar;280(3):G368-80. doi: 10.1152/ajpgi.2001.280.3.G368. PMID 11171619
- [Result] Dimidi E, Christodoulides S, Fragkos KC, Scott SM, Whelan K. The effect of probiotics on functional constipation in adults: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2014 Oct;100(4):1075-84. doi: 10.3945/ajcn.114.089151. Epub 2014 Aug 6. PMID 25099542
- [Result] Koebnick C, Wagner I, Leitzmann P, Stern U, Zunft HJ. Probiotic beverage containing Lactobacillus casei Shirota improves gastrointestinal symptoms in patients with chronic constipation. Can J Gastroenterol. 2003 Nov;17(11):655-9. doi: 10.1155/2003/654907. PMID 14631461